CLINICAL TRIAL: NCT06182917
Title: A Study for Assessing the Value of Minimal Residual Disease Detection in Disease Monitoring of CA125 Non-sensitive Ovarian Cancer Patients
Brief Title: Prognostic Value of MRD Detection in CA125 Non-sensitive Ovarian Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Rutie Yin, West China Second University Hospital, West China Second University Hospital
Other Study IDs: WCSUH20231108
Record Dates: First submitted 2023-11-25; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ctDNA alternation during the treatment of Ovarian cancer: Tumor samples of included patients were detected by WES, and 16 major clonal mutation sites were screened for the personalized monitoring panel. All patients received blood ctDNA detection to monitor the major clonal alternation after 3 cycels treatment or 3 months after therapy, at the same time, the detection of serum tumor markers (CA125) and imaging examination were carried out, in order to evaluate the MRD detection efficiency.

SUMMARY:
Ovarian cancer ranks third in the incidence of gynecologic malignancies, while mortality ranks first. The tumor marker CA125 is the most concerned tumor marker in the clinical monitoring prognosis of ovarian cancer, and an elevated CA125 indicates a later stage and a worse prognosis. However about 20% of patients with ovarian cancer have low CA125 expression. Therefore, CA125 is not sensitive to some ovarian cancers with a high risk of recurrence. How to improve the diagnostic performance of these CA125-insensitive patients is a difficult problem in current research. Minimal residual disease (MRD) refers to the residual tumor components in the body of tumor patients after achieving complete remission through treatment. MRD detection is mainly achieved by liquid biopsy, and residual tumor components can be detected by circulating tumor DNA (ctDNA). This study aims to explore the value of MRD (ctDNA) in the risk assessment of CA125 non sensitive ovarian cancer populations by combining ctDNA with traditional imaging and serological tumor markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* Pathologically confirmed ovarian cancer;
* CA125 ≤200U/ml at first diagnosis or recurrence;
* Physical condition score PS ≤ 2 points;
* Enough tumor samples for WES detection;
* Patients and their families can understand and are willing to participate in this study and provide written informed consent.

Exclusion Criteria:

* Patients unable to provide sufficient tissue / blood samples for research detection;
* Pregnant or lactating women;
* Other diseases considered by the research doctor to affect the prognosis and survival;

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: This study intends to include 35 patients with low CA125 level ovarian cancer at first diagnosis or recurrence between the ages of 18-75 years old.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The prognostic value of MRD | 12 months
  The sensitivity of MRD in CA125 low level ovarian patients.

SECONDARY OUTCOMES:
Progress Free Survival | From date of the beginning of therapy to disease metastasis or recurrence due to any cause,assessed up to 24 months
  PFS differences in patients with different MRD level

CONTACTS AND LOCATIONS:
Overall Officials: Mengpei Zhang, Principal Investigator — West China Second University Hospital; Rui Li, Principal Investigator — West China Second University Hospital
Locations (1):
- west china second University， SICHUAN University, China, Chengdu, Sichuan, China